CLINICAL TRIAL: NCT02106065
Title: Dementia Caregiver Rehabilitation: Enhancing Veteran and Family-Centered Care
Brief Title: VA Cultivating Access to Resources, Education, and Skills for Dementia Caregivers
Acronym: VACARES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E1240-W; 5IK2RX001240-02 (NIH)
Record Dates: First submitted 2014-03-27; First posted 2014-04-07 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Dementia; Caregivers; Neurodegenerative Diseases; Brain Diseases
Keywords: Dementia; Caregivers; Neurodegenerative Diseases; Brain Diseases; Cost of Illness; Stress, Psychological; Depression; Vital Statistics; Mortality; Behavioral Symptoms; Residential Facilities; Emergency Medical Services; Long-Term Care
MeSH Terms: conditions — Dementia; Neurodegenerative Diseases; Brain Diseases; Stress, Psychological; Depression; Behavioral Symptoms | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- In-person Education and Skill-Building Rehabilitation (ESBR-i) Condition (Experimental): Education and Skill-Building Rehabilitation delivered in clinic
  Interventions: Behavioral: Education and Skill-Building Rehabilitation (ESBR)
- Education and Skill-Building Rehabilitation over Video (ESBR-V) Condition (Experimental): Education and Skill-Building Rehabilitation delivered via video telehealth.
  Interventions: Behavioral: Education and Skill-Building Rehabilitation (ESBR)
- Usual Care Condition (Active Comparator): Usual Care plus supplemental paper education materials
  Interventions: Other: Supplemental Education Materials

INTERVENTIONS:
Behavioral: Education and Skill-Building Rehabilitation (ESBR) — ESBR intervention consists of four, 90-minute sessions over a 4-6 week period. These four sessions are supplemented with booster sessions at 3 and 9 months post-intervention. Each group session (10 or fewer participants) is attended either in-clinic or via video telehealth technology within the VAPAHCS.
  Other Names: ESBR
  Arms: Education and Skill-Building Rehabilitation over Video (ESBR-V) Condition; In-person Education and Skill-Building Rehabilitation (ESBR-i) Condition
Other: Supplemental Education Materials — Participants randomized to the Usual Care (UC) group will receive supplemental educational materials related to aging and dementia.
  Arms: Usual Care Condition

SUMMARY:
The purpose of this study is to study the effects of an education and skill-building intervention on family caregivers of Veterans with dementia.

DETAILED DESCRIPTION:
According to VA estimates, nearly 500,000 Veterans suffer from dementia. There is currently no cure for dementia. Ultimately, dementia will have a large impact on quality of life in Veterans and families, lead to expensive nursing home placement, and decrease life expectancy for patients and family caregivers. The experience of high burden in a caregiver for a Veteran with dementia increases the likelihood of permanent nursing home placement and can separate Veterans from their families. To address the high burden of caring for a Veteran with dementia, the investigators aim to study the effect of a rehabilitative intervention for family caregivers of Veterans with dementia. This novel approach will use video technology that can reach caregivers in rural areas who do not have easy access to major VA medical centers.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria -- Participants must:

* be adults (age 18)
* report distress associated with being the primary caregiver for a Veteran family member with all-cause dementia
* reporting at least 2 of the following 6 items at baseline assessment: felt overwhelmed, felt like they often needed to cry, were angry or frustrated, felt they were cut off from family or friends, reported moderate to high levels of general stress, or felt their health had declined
* provide at least one hour of care (supervision or direct assistance) per week over the past 3 months (other sources of caregiving for the Veteran with dementia can also be utilized; e.g., respite, home health aide, other family members, etc.)
* be proficient in spoken and written English
* be capable of providing informed consent

Exclusion Criteria:

Exclusion criteria -- Potential participants will be screened and excluded for:

* current or lifetime history of any psychiatric disorder with psychotic features
* prominent suicidal or homicidal ideation
* having met DSM-IV criteria for drug or alcohol abuse or dependence (except nicotine) within the past six months
* presence of alcohol intoxication (by breathalyzer) or alcohol withdrawal (by exam) during study recruitment or participation
* diagnosis of probable or possible dementia
* a Telephone Cognitive Screen score of < 20
* participation in another caregiver intervention within the past year
* lack of regular access to a telephone
* illness that would prevent 24 months of study participation
* planned transfer of care receiver to another caregiver or nursing home within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-02-21 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blake K Scanlon, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA; Jennifer K Fairchild, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ESBR-i: Education and Skill-Building Rehabilitation (in-clinic)
  Education and Skill-Building Rehabilitation (ESBR): ESBR intervention consists of four, 90-minute sessions over a 4-6 week period. These four sessions are supplemented with booster sessions at 3 and 9 months post-intervention. Each group session (10 or fewer participants) is attended either in-clinic or via video telehealth technology within the VAPAHCS.
- ESBR-v: Education and Skill-Building Rehabilitation (over video telehealth)
  Education and Skill-Building Rehabilitation (ESBR): ESBR intervention consists of four, 90-minute sessions over a 4-6 week period. These four sessions are supplemented with booster sessions at 3 and 9 months post-intervention. Each group session (10 or fewer participants) is attended either in-clinic or via video telehealth technology within the VAPAHCS.
- Usual Care: Usual Care plus supplemental paper education materials
  Supplemental Education Materials: Participants randomized to the Usual Care (UC) group will receive supplemental educational materials related to aging and dementia.
Period: Overall Study
Arm/Group | ESBR-i | ESBR-v | Usual Care
Started | 6 | 11 | 15
6 Month Completion | 3 | 8 | 5
Completed | 3 | 8 | 5
Not Completed | 3 | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ESBR-i | ESBR-v | Usual Care | Total
Number analyzed (Participants) | 6 | 11 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (7.0) | 69.8 (10.7) | 65 (10.9) | 68.6 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 14 | 22
  Male | 0 | 9 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 1 | 6
  White | 2 | 8 | 10 | 20
  More than one race | 1 | 0 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 1 | 1
Zarit Burden Inventory [Mean (Standard Deviation); unit: units on a scale] — The Zarit Burden Inventory is a self-report measure of caregiver burden. Scores range from 0-88 with higher scores indicating more severe burden.
  units on a scale | 50.0 (5.2) | 30.6 (12.5) | 40.8 (12.0) | 40.47 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: Zarit Burden Inventory
Description: The Zarit Burden Inventory is a self-report measure of caregiver burden. Higher scores on this assessment indicate greater levels of caregiver burden. Potential scores range from 0-88 with higher scores indicating more severe burden.
Time Frame: change from baseline at 6-months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESBR-i | ESBR-v | Usual Care
Number analyzed (Participants) | 3 | 8 | 5
score on a scale | 2.0 (2.6) | -0.4 (5.0) | 1.6 (3.0)

2. Secondary Outcome: Center for Epidemiological Studies-Depression
Description: change in caregiver depressive symptoms as measured by the Center for Epidemiological Studies-Depression (CES-D). Scores on the CES-D can range from 0-60 with higher scores suggesting greater depressive symptomatology.
Time Frame: change from baseline at 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESBR-i | ESBR-v | Usual Care
Number analyzed (Participants) | 3 | 8 | 5
score on a scale | 2.0 (6.9) | 0.1 (3.3) | -0.2 (5.3)

3. Secondary Outcome: Long-term Care Placement Status (Care Recipient)
Description: Based on caregiver interview, permanent placement of the care recipient in LTC will be ascertained
Time Frame: 6-months post intervention
Population: This data was not collected thus is not reported here.
Arm/Group | ESBR-i | ESBR-v | Usual Care
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change in All-cause Mortality Status (Care Recipient)
Description: Based on caregiver interview, care recipient mortality status will be ascertained
Time Frame: 6-months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | ESBR-i | ESBR-v | Usual Care
Number analyzed (Participants) | 3 | 8 | 5
Participants | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: 24 Months
Arm/Group | ESBR-i | ESBR-v | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/6 | 0/11 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/11 | 0/15
Other Adverse Events (participants affected / at risk) | 0/6 | 0/11 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ESBR-i (N=6) | ESBR-v (N=11) | Usual Care (N=15)
Musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT02106065/Prot_SAP_000.pdf